CLINICAL TRIAL: NCT00180622
Title: Non-Invasive Markers for Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Markers for Chronic Obstructive Pulmonary Disease (COPD)
Status: Withdrawn | Type: Observational
Why Stopped: No resources available
Sponsor: Imperial College London (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: SD-000-068
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Healthy Non-smokers; Current Smokers; COPD Patients
MeSH Terms: interventions — Carbon Monoxide; Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Spirometry
Procedure: Exhaled Nitric Oxide and Carbon Monoxide
Procedure: Exhaled Breath Condensate
Procedure: Induced Sputum
Procedure: CT Scan
Procedure: Blood test
Procedure: St Georges Questionnaire
Procedure: Bodypletysmography

SUMMARY:
The primary aim of this study is to exploit a difference between COPD patients, chronic smokers without COPD and healthy non-smoking subjects. This will help to assess the utility of inflammatory and oxidative markers in exhaled air and sputum and to compare them with the lung function, clinical parameters and computerised tomography (CT).

ELIGIBILITY:
Inclusion Criteria:

Healthy non-smokers

* FEV1 >80% predicted
* FEV1 reversibility of <10% after inhaled (beta2-agonists

Current smokers

* FEV1 no less than 80% predicted
* FEV1 reversibility of <10% after inhaled (beta2-agonists
* Smoking history of > 10 pack-years

Moderate COPD

* FEV1 40-59% predicted
* FEV1 reversibility of <10% after inhaled (beta2-agonists
* Smoking history of > 10 pack-years**

Severe COPD

* FEV1 <40% predicted
* FEV1 reversibility of <10% after inhaled (beta2-agonists
* Smoking history of > 10 pack-years

Exclusion Criteria:

* FEV1 increases by 200 ml and 15% of the baseline value after inhaled (beta2-agonists
* Asthma
* unstable disease (FEV1 <35% predicted) and/or current, or within the last 4 weeks, respiratory tract infection.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2001-07-01 (Estimated); Primary Completion 2002-07-01 (Estimated); Study Completion 2002-07-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sergei A Kharitonov, MD PhD, Principal Investigator — Imperial College London; Peter J Barnes, MA DM DSc FRCP, Principal Investigator — Imperial College London
Locations (1):
- Section of Airway Disease, Asthma Lab, Imperial College London, Royal Brompton Hospital, London, United Kingdom